CLINICAL TRIAL: NCT05320796
Title: The Bioavailability and Effect on Pouch pH of Esomeprazole as Tablets or in Solution After Laparoscopic Proximal RYGB for Morbid Obesity - an Investigator Blinded Pilot Study
Brief Title: The Bioavailability and Effect on Pouch pH of Esomeprazole After Gastric Bypass
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prof Urs Zingg (Other)
Responsible Party: Sponsor-Investigator, Prof Urs Zingg, Prof. Dr., Spital Limmattal Schlieren
Organization: Spital Limmattal Schlieren (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LS-202112
Record Dates: First submitted 2021-12-29; First posted 2022-04-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Gastric Reflux; Ulcer, Gastric
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux; Stomach Ulcer | interventions — Gastroscopy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Esomeprazol administered in tablets (Esomeprazol MUT Sandoz® 40mg) ¨ or in solution (Esomeprazol MUT Sandoz® 40mg in 10ml tap water)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Solution (Experimental): Esomeprazol MUT Sandoz® 40mg as a single dose will be dissolved in 10ml tap water to create a solution and then applied per oral
  Interventions: Diagnostic Test: upper endoscopy
- Tablet (Active Comparator): Esomeprazo MUT Sandozl® 40mg tablet as a single dose will be given orally
  Interventions: Diagnostic Test: upper endoscopy

INTERVENTIONS:
Diagnostic Test: upper endoscopy — A wireless BRAVO™ - pH monitoring device is placed and the participant is discharged with ongoing pH monitoring. The next day, the participant is randomized to either receive Esomeprazol MUT Sandoz® tablet 40mg or Esomeprazol MUT Sandoz® 40mg in solution. Serum concentration of Esomeprazol is measured at 0, 60 and 120 minutes and the patient is discharged after. After 48 hours of pH monitoring, the patient returns the BRAVO™ - recorder, adverse events are assessed and the study is terminated.
  Other Names: blood sample

SUMMARY:
The objective of this study is to investigate the effect of Esomeprazol administered in tablets (Esomeprazol MUT Sandoz® 40mg) or in solution (Esomeprazol MUT Sandoz® 40mg in 10ml tap water) on acid production in the gastric pouch by measuring the intragastric pH and the serum concentration of esomeprazole.

DETAILED DESCRIPTION:
To assess the clinical effect of the esomeprazole absorption after Roux-en-Y gastric bypass, we intend to measure the serum concentration after administration as intact capsules or open in solution and correlate it with the pH in the gastric pouch, measured with the wireless BRAVOTM capsule pH measurement system. The feasibility and safety of the wireless pH monitoring system has been shown before.

The patients who met all the inclusion criteria undergo a routine upper endoscopy one year after RYGB. At the end of the endoscopy, the wireless BRAVO™ - pH monitoring device is placed and the participant is discharged with ongoing pH monitoring. The next day, the participant is randomized to either receive Esomeprazol MUT Sandoz® tablet 40mg or Esomeprazol MUT Sandoz® 40mg in solution. Serum concentration of Esomeprazol is measured at 0, 60 and 120 minutes and the patient is discharged after. After 48 hours of pH monitoring, the patient returns the BRAVO™ - recorder, adverse events are assessed and the study is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Proximal Roux-en-Y gastric bypass with linear stapled anastomosis 12 months prior to the study investigation
* Routine administration of proton pump inhibitors for 6 months postoperatively
* No intake of proton pump inhibitors at least 4 weeks prior to study investigation
* No marginal ulcers in upper endoscopy prior to placement of wireless BRAVO™ pH monitoring capsule
* No symptoms related to gastro-esophageal reflux or marginal ulcers (i.e. epigastric pain, retrosternal burning, regurgitation)
* Informed consent as documented by signature

Exclusion Criteria:

* Known intolerance or allergy for Esomeprazol
* Contraindication for upper endoscopy
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Women who are pregnant or breast feeding Major hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pH | 48 hours
  The primary outcome is the total time, in which the pH in the gastric pouch is <4 measured with wireless BRAVO™ - pH monitoring.

SECONDARY OUTCOMES:
serum concentration | 2 hours after administration
  The main secondary outcome is the serum concentration of Esomeprazol in nanogramm per mililiter in the blood serum at 0, 60 and 120 minutes after drug administration either as tablet or in solution.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, Prof., Principal Investigator — Limmattal Hospital
Locations (1):
- Spital Limmattal, Schlieren, Switzerland

IPD SHARING:
Plan to Share IPD: No